CLINICAL TRIAL: NCT02665858
Title: OCT Imaging of Papilledema in Pediatric Idiopathic Intracranial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0035-15-HYMC
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Pediatric Idiopathic Intracranial Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IIH Patients (Active Comparator): Patients diagnosed with Idiopathic Intracranial Hypertension who undergo OCT imaging
  Interventions: Other: OCT Imaging
- Control Group (Active Comparator): Patients diagnosed with headache with ruled out Idiopathic Intracranial Hypertension who undergo OCT imaging
  Interventions: Other: OCT Imaging

INTERVENTIONS:
Other: OCT Imaging

SUMMARY:
Longitudinal clinical observation of optic nerve head, using slit lamp fundoscopy, guides therapy in pediatric idiopathic intracranial hypertension (IIH) patients; however, it remains a limited method of producing quantitative data in evaluating in patients with IIH.

In this study we intend to compare, by using spectral domain optical coherence tomography (OCT), the mean retinal nerve fiber layer thickness and total retinal thickness (RNFLT/TRT) of the optic nerve of newly diagnosed IIH children to a control group. This will provide a quantitative measure for follow-up and treatment of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Children with suspected IIH

Exclusion Criteria:

* Retinal disease
* High refractive error
* Unable to undergo OCT imaging

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of RNFLT/TRT Thickness | One year

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Cohen, MD, PhD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No